CLINICAL TRIAL: NCT06948968
Title: Turkish Version of the Adapted Social Role Participation Questionnaire for Ankylosing Spondylitis: A Study on Its Validity and Reliability
Brief Title: Turkish Version of the Adapted Social Role Participation Questionnaire
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tugba Gokbel, Assistant Prof Dr, Kocaeli University
Other Study IDs: 6/56
Record Dates: First submitted 2025-03-12; First posted 2025-04-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Ankylosing Spondylitis; Participation, Patient
Keywords: Ankylosing Spondylitis; Participation; Social Role Participation; SRPQ; Turkish Adaptation
MeSH Terms: conditions — Spondylitis, Ankylosing; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Social Role Participation Questionnaire — Validity and Reliability of the Turkish Version of the Adapted Social Role Participation Questionnaire in Ankylosing Spondylitis

SUMMARY:
Participation, as defined by the International Classification of Functioning, Disability, and Health (ICF), refers to "engagement in a life situation" and is a key component of functional health beyond physical impairments or activity limitations. Social role participation encompasses various aspects of life, including work, family commitments, social interactions, and leisure activities.

Ankylosing Spondylitis (AS), a chronic inflammatory disease affecting the axial skeleton, significantly impacts patients' ability to maintain social roles due to pain, stiffness, and reduced mobility. Existing studies highlight limitations in employment, relationships, education, and leisure activities among AS patients. While various scales assess participation, the Social Role Participation Questionnaire (SRPQ) uniquely emphasizes subjective aspects such as role importance and satisfaction with performance.

Although validated versions of the SRPQ exist in English, Dutch, and Chinese populations, no culturally adapted tool is available for Turkish-speaking AS patients. This study aims to translate the SRPQ into Turkish and evaluate its validity and reliability as a culturally appropriate instrument for assessing social role participation.

DETAILED DESCRIPTION:
The International Classification of Functioning, Disability and Health (ICF) defines participation as "engagement in a life situation" viewing the concept of participation that a functional element beyond body functions and activity limitations. Role participation can be considered in a multifaceted manner. This includes not only participation in a role but but also perceptions of the role's importance, the assessment of limitations or challenges in-role performance, and satisfaction with the individual's ability to fulfill a role according to personal preference. Social role participation encompasses various aspects of an individual's life, including work, family commitments, social interactions, and leisure activities.

Ankylosing Spondylitis (AS), with its chronic, inflammatory, and progressive nature, primarily affects the sacroiliac joints and axial skeleton, leading to pain, joint stiffness, and reduced spinal mobility in individuals. Peripheral and extra-articular symptoms may also occur. Consequently, the physical function loss that develops in individuals reduces their quality of life and productivity, negatively impacting social role participation and the ability to maintain communal roles, affecting their overall well-being. According to the literature, it is documented that individuals with AS experience mild or greater limitations in areas such as recreation and leisure, social life, employment, close relationships, formal and informal social relationships, basic and complex interpersonal interactions, family relationships, education, and contributing to others' well-being.

Existing scales related to participation differ based on the roles they include and the social dimensions they asses (vary based on the different participation roles they include and the dimensions of social roles they measure). Unlike other participation scales that assess social role participation based on frequency, restriction, or role occupation, the SRPQ is a promising tool that emphasizes the assessment of an individual's subjective aspects, particularly their desires and satisfactions, across a wide range of roles in various dimensions. From an individual perspective, the "satisfaction" dimension is particularly noteworthy, as it can be linked to numerous aspects of participation performance and other qualitative dimensions. It provides additional insights into the personal assessment of role performance. Furthermore, the "importance of the role" dimension, which reflects the value an individual assigned to a role, serves as a potential factor that qualifies performance scores. Its direct assessment may offer a possible approach to studying response shift phenomena, which influence many of the subjective aspects of participation.

The English, Dutch, and Chinese versions of the SRPQ have been proven to be reliable and valid tools for measurement assessing social role participation in individuals with AS. Davis et al. have reported that this tool can also be used to evaluate the complex relationships between symptoms, disability, and participation, along with the personal and environmental contextual factors that influence them.

Currently, in Turkey, there is no valid and reliable tool that simultaneously evaluates the importance, physical difficulty, and satisfaction related to social role participation in individuals with AS. This study aims to translate the SRPQ, into Turkish as it encompasses all dimensions of social role participation, and to evaluate its validity and reliability among Turkish-speaking individuals with AS, thereby providing a culturally appropriate assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AS according to the modified New York criteria
* Being over 18 years old
* To comprehend Turkish and communicate fluently in the Turkish language

Exclusion Criteria:

* Having severe psychiatric conditions
* Concomitant severe medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Reliability of the Turkish Version of the Adapted Social Role Participation Questionnaire (SRPQ) in Ankylosing Spondylitis | 2018-2022
  To assess reliability, the Social Role Participation Questionnaire (SRPQ) was completed twice by the same participants in a quiet room at two-week intervals. Internal consistency was evaluated using Cronbach's alpha (α ≥ 0.70, acceptable), and test-retest reliability was assessed using the Intraclass Correlation Coefficient (ICC ≥ 0.85, excellent), based on a two-way mixed-effects model with absolute agreement. The SRPQ includes three dimensions: Role Importance (1-5), Satisfaction with Performance (1-5), and Physical Difficulty (1-4). Higher scores on Role Importance and Satisfaction indicate better perceived participation, while higher scores on Physical Difficulty reflect greater difficulty in performing roles.
Validity of the Turkish Version of the Adapted Social Role Participation Questionnaire (SRPQ) in Ankylosing Spondylitis | 2018-2022
  Construct validity was evaluated by correlating SRPQ scores with three validated instruments: the Ankylosing Spondylitis Quality of Life Scale (ASQoL), Short Form-36 Health Survey (SF-36), and Work Productivity and Activity Impairment Questionnaire (WPAI). ASQoL (0-18) assesses disease-specific quality of life, with higher scores reflecting greater impairment. SF-36 covers eight health domains (0-100), with higher scores indicating better health. Participation was captured in the social functioning, role-physical, and role-emotional domains. The WPAI (0-100%) measures work productivity and activity impairment over the prior week, with higher percentages indicating greater disability. Spearman correlation coefficients were used and interpreted as poor (<0.20), fair (0.21-0.40), moderate (0.41-0.60), very good (0.61-0.80), or excellent (>0.81). The scoring directionality of each scale supports the interpretation of SRPQ's convergent and discriminant validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jimenez Bunuales MT, Gonzalez Diego P, Martin Moreno JM. [International classification of functioning, disability and health (ICF) 2001]. Rev Esp Salud Publica. 2002 Jul-Aug;76(4):271-9. doi: 10.1590/s1135-57272002000400002. Spanish. PMID 12216167
- [Background] Davis AM, Palaganas MP, Badley EM, Gladman DD, Inman RD, Gignac MA. Measuring participation in people with spondyloarthritis using the social role participation questionnaire. Ann Rheum Dis. 2011 Oct;70(10):1765-9. doi: 10.1136/ard.2010.149211. Epub 2011 Jul 25. PMID 21791450
- [Background] Sieper J, Braun J, Rudwaleit M, Boonen A, Zink A. Ankylosing spondylitis: an overview. Ann Rheum Dis. 2002 Dec;61 Suppl 3(Suppl 3):iii8-18. doi: 10.1136/ard.61.suppl_3.iii8. PMID 12381506
- [Background] van Echteld I, Cieza A, Boonen A, Stucki G, Zochling J, Braun J, van der Heijde D. Identification of the most common problems by patients with ankylosing spondylitis using the international classification of functioning, disability and health. J Rheumatol. 2006 Dec;33(12):2475-83. Epub 2006 Oct 15. PMID 17013999
- [Background] Gignac MA, Backman CL, Davis AM, Lacaille D, Mattison CA, Montie P, Badley EM. Understanding social role participation: what matters to people with arthritis? J Rheumatol. 2008 Aug;35(8):1655-63. Epub 2008 Jun 15. PMID 18597401
- [Background] Dijkers MP. Issues in the conceptualization and measurement of participation: an overview. Arch Phys Med Rehabil. 2010 Sep;91(9 Suppl):S5-16. doi: 10.1016/j.apmr.2009.10.036. PMID 20801280
- [Background] van Genderen S, Plasqui G, Lacaille D, Arends S, van Gaalen F, van der Heijde D, Heuft L, Keszei A, Luime J, Spoorenberg A, Landewe R, Gignac M, Boonen A. Social Role Participation Questionnaire for patients with ankylosing spondylitis: translation into Dutch, reliability and construct validity. RMD Open. 2016 Feb 1;2(1):e000177. doi: 10.1136/rmdopen-2015-000177. eCollection 2016. PMID 26870393
- [Background] Zhang G, Li J, Liu D, Wang T, Wang Y, Xu W. Translation and validation of the Chinese Social Role Participation Questionnaire in patients with ankylosing spondylitis. Clin Rheumatol. 2018 Mar;37(3):655-660. doi: 10.1007/s10067-017-3915-z. Epub 2017 Nov 18. PMID 29151172
- See also: International classification of functioning, disability and health (ICF) 2001 — https://pubmed.ncbi.nlm.nih.gov/12216167/
- See also: Measuring participation in people with spondyloarthritis using the social role participation questionnaire — https://pubmed.ncbi.nlm.nih.gov/21791450/
- See also: Ankylosing spondylitis: an overview — https://pubmed.ncbi.nlm.nih.gov/12381506/
- See also: Identification of the most common problems by patients with ankylosing spondylitis using the international classification of functioning, disability and health — https://pubmed.ncbi.nlm.nih.gov/17013999/
- See also: Understanding social role participation: what matters to people with arthritis? — https://pubmed.ncbi.nlm.nih.gov/18597401/
- See also: Issues in the conceptualization and measurement of participation: an overview — https://pubmed.ncbi.nlm.nih.gov/20801280/
- See also: Social Role Participation Questionnaire for patients with ankylosing spondylitis: translation into Dutch, reliability and construct validity — https://pubmed.ncbi.nlm.nih.gov/26870393/
- See also: Translation and validation of the Chinese Social Role Participation Questionnaire in patients with ankylosing spondylitis — https://pubmed.ncbi.nlm.nih.gov/29151172/